CLINICAL TRIAL: NCT00003017
Title: Phase II Clinical Trial of Interleukin-12 in Patients With Advanced, Recurrent or Inoperable Carcinoma of the Cervix
Brief Title: Interleukin-12 in Treating Patients With Advanced or Recurrent Cancer of the Cervix
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065597; ECOG-E1E96
Record Dates: First submitted 1999-11-01; First posted 2004-04-22 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2004-07

CONDITIONS: Cervical Cancer
Keywords: stage IV cervical cancer; recurrent cervical cancer; cervical squamous cell carcinoma; cervical adenocarcinoma; cervical adenosquamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Interleukin-12 Subunit p35

INTERVENTIONS:
Biological: recombinant interleukin-12

SUMMARY:
RATIONALE: Interleukin-12 may kill tumor cells by stopping blood flow to the tumor and by stimulating a person's white blood cells to kill cancer cells in the cervix.

PURPOSE: Phase II trial to study the effectiveness of interleukin-12 in treating patients who have advanced or recurrent cancer of the cervix.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rates, duration of response, and survival in women with advanced, recurrent, or inoperable cervical cancer treated with interleukin-12. II. Determine the toxic effects of systemic interleukin-12 in these patients. III. Correlate response to therapy and survival with the presence or absence of human papilloma virus (HPV), and the specific subtype of HPV, in these patients.

OUTLINE: Patients are stratified according to prior chemotherapy (yes vs no). Patients receive induction interleukin-12 IV over 5-20 seconds on day -13 and then daily on days 1-5. Treatment continues every 21 days in the absence of unacceptable toxicity or disease progression. Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 78 patients (39 per stratum) will be accrued for this study within 26 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven stage IV or recurrent squamous cell, adenosquamous, or adenocarcinoma of the uterine cervix including: Lung, liver, lymph node, or skin metastases OR Retroperitoneal disease OR Other advanced measurable disease OR Positive paraaortic lymph nodes Measurable disease that is beyond the scope of conventional radiation therapy or surgery, or recurrent after radiation therapy or surgery Measurable, recurrent disease within a previously irradiated field must have increased in size by 100% on at least 2 successive scans, MRI, or physical examinations

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 OR Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times the upper limit of normal (ULN) AST and ALT no greater than 2 times ULN Renal: Creatinine no greater than 2.0 mg/dL Creatinine clearance at least 60 mL/min Cardiovascular: No New York Heart Association class III/IV heart disease No uncontrolled congestive heart failure or angina Pulmonary: No chronic obstructive pulmonary disease Gastrointestinal: No evidence of active gastrointestinal bleeding No active peptic ulcer disease No inflammatory bowel disease Other: Normal diet required No known active infections HIV negative AIDS-related complex (ARC) negative No substance abuse or psychiatric problems No evidence of autoimmune disease No other prior invasive malignancy except resected basal cell or squamous cell skin cancer Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: 1 prior biologic therapy allowed At least 4 weeks since prior biologic therapy Chemotherapy: 1 prior adjuvant chemotherapy regimen allowed 1 prior chemotherapy regimen for advanced disease allowed At least 4 weeks since prior chemotherapy No concurrent chemotherapy Endocrine therapy: No concurrent steroid therapy No concurrent megestrol acetate Radiotherapy: See Disease Characteristics No concurrent radiotherapy Surgery: See Disease Characteristics At least 2 weeks since prior surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-07; Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Wadler, MD, Study Chair — Albert Einstein College of Medicine
Locations (9):
- United States (9):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Hunterdon Regional Cancer Center, Flemington, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Vanderbilt Cancer Center, Nashville, Tennessee

REFERENCES:
- [Result] Wadler S, Levy D, Frederickson HL, Falkson CI, Wang Y, Weller E, Burk R, Ho G, Kadish AS; Eastern Cooperative Oncology Group. A phase II trial of interleukin-12 in patients with advanced cervical cancer: clinical and immunologic correlates. Eastern Cooperative Oncology Group study E1E96. Gynecol Oncol. 2004 Mar;92(3):957-64. doi: 10.1016/j.ygyno.2003.12.022. PMID 14984966